CLINICAL TRIAL: NCT06734325
Title: Effectiveness of Mobile Oral Health Intervention on Oral Hygiene and Oral Health Literacy Among Orthodontic Patients: a Randomized Controlled Clinical Trial)
Brief Title: Mobile Oral Health Intervention Effectiveness on Orthodontic Patients' Oral Hygiene and Oral Health Literacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nermine Balbaa, Teaching assistant, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0913-05/2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Oral Health Literacy; Oral Hygiene
Keywords: oral health literacy; oral hygiene; orthodontic patients; mobile oral health intervention; whatsapp; messages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Oral Health Intervention (Experimental): Mobile oral health intervention in addition to oral hygiene instructions
  Interventions: Behavioral: Mobile Oral Health Intervention
- Control (No Intervention): oral hygiene instructions only

INTERVENTIONS:
Behavioral: Mobile Oral Health Intervention — 46 messages delivered over a 3-month period (12 weeks) via WhatsApp
  Arms: Mobile Oral Health Intervention

SUMMARY:
Orthodontic patients face unique challenges in maintaining optimal oral hygiene due to the presence of fixed orthodontic appliances, which tend to increase plaque retention, leading to gingival inflammation. Oral Health Literacy (OHL) plays a role in an individual's ability to understand and implement oral hygiene instructions effectively. Mobile oral health interventions involve the use of mobile technology such as smartphones to improve oral hygiene practices and outcomes.

Aim of the study: To assess the effectiveness of a mobile oral health intervention using WhatsApp messages as compared to standard oral hygiene instructions on oral hygiene status and OHL level among orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing orthodontic treatment with fixed appliances in both arches for the first time.
2. Patients between the age of 16 and 25 years.
3. Participants must own a smartphone with WhatsApp installed.
4. Those who agree to be part of the research project and accept the informed consent.

Exclusion Criteria:

1. The presence of systemic diseases affecting oral health.
2. Patients with cleft lip and/or palate.
3. Functional and orthognathic patients.
4. Previous orthodontic treatment.
5. Patients with a removable appliance.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Oral Health Literacy | Change from baseline to 1 month, 3 months, 6 months
  oral health literacy as measured by the Oral Health Literacy - Adult Questionnaire (OHL-AQ). Scores of all questions answered by participants will be added to obtain the overall score of OHL ranging from 0 to 17. Scores are categorized into three groups: Inadequate (0-9), Borderline (10-11), and Adequate (12-17) OHL level

SECONDARY OUTCOMES:
Oral Hygiene | Change from baseline to 1 month, 3 months, 6 months
  assessed by the Silness-Löe Plaque Index (PI) to provide mean PI score for each tooth ranging from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Nermine Balbaa, BDS, Principal Investigator — Teaching Assistant, Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Pubalan S, Zi Hong O, Yongxian T, Mabel L. Assessing effectiveness of WhatsApp messaging program in oral hygiene care for orthodontic patients: A randomised controlled trial. J Orthod. 2024 Dec;51(4):407-414. doi: 10.1177/14653125241230561. Epub 2024 Feb 17. PMID 38366912
- [Background] Cho HA, Im AJ, Sim YR, Jang HB, Lim HJ. The association between oral health literacy and oral health behaviors in North Korean defectors: a cross-sectional study. BMC Public Health. 2020 Jul 7;20(1):1074. doi: 10.1186/s12889-020-08550-7. PMID 32635907
- [Derived] Balbaa NM, Hamza MA, Abdelaziz WE, Adham MM. Effectiveness of mobile oral health intervention on orthodontic patients' oral hygiene and oral health literacy: a randomised controlled clinical trial. BMC Oral Health. 2025 Dec 12;26(1):113. doi: 10.1186/s12903-025-07423-y. PMID 41382113